CLINICAL TRIAL: NCT06999239
Title: Evaluation of the Effect of Laser Therapy on Lateral Pterygoid Muscle in Patients With Wilke's Stage I and II Temporomandibular Disorders (TMD): Case Series Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aliaa ibrahim fathy, doctor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Treatment of TMD by laser
Record Dates: First submitted 2025-05-09; First posted 2025-05-31 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Laser; Temporomandibular Joint Disorders; Lateral Pterygoid Muscle
Keywords: laser therapy, lateral pterygoid muscle, Wilke's, stage I and II, TMD.
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Laser Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one arm(case series0 (Experimental)
  Interventions: Procedure: laser therapy in TMD

INTERVENTIONS:
Procedure: laser therapy in TMD — In this study patients will receive the Low-level laser therapy with a 635 nm wavelength diode laser (Lasotronix, Diode Laser DiodeLX model SMART M; Zytnia, Piaseczno, Poland) with 200 mW in a continuous mode, using a handpiece with a cylindrical applicator with a diameter of 8 mm in contact mode extra-orally, fiber-optic applicator with a diameter of 8 mm in contact mode intraorally, with a power density of 400 mW/cm2, delivering 10-12 J/cm2 on each application point, over a period of 20 sec.
  There are two methods for examination of lateral pterygoid muscle: digital palpation and functional manipulation.
  For digital palpation of lateral pterygoid muscle, we place our index finger or tip of our little finger in the vestibular area adjacent to the maxillary third molar.
  Functional manipulation of the inferior head of lateral pterygoid muscle: It is best accomplished by having the patient make a protrusive movement against resistance to contract it since this muscle is the primary pro

SUMMARY:
The purpose of this study will be to evaluate the effect of laser therapy on lateral pterygoid muscle in patients with Wilke's stage I and II temporomandibular disorders (TMD).

ELIGIBILITY:
Inclusion criteria:

1. Patients age between 16-50 years with no sex predilection.
2. Patients who will be free from any systemic diseases that affect temporomandibular joint.
3. Patients who will be diagnosed with wilk's stage I and II temporomandibular disorders (TMD).
4. Patients who will be ready to give informed consent.

Exclusion Criteria:

1. Patients with previous temporo-mandibular surgeries.
2. Patients with previous facial fracture.
3. Patients who will be under another type of treatment for TMD (e.g., occlusal splints, pharmacological drugs, or head and neck surgery).
4. Patients who will not attend the proposed treatment sessions or follow-up visits.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pain: will be obtained by Visual analogue scale (VAS). | pain will be measured : 1.day1 before the start of laser therapy, 2.week 1 3. week2 4.week 3 5. week 4 6.one month later 7. 3 months later.
  Pain: will be obtained by Visual analogue scale (VAS).

SECONDARY OUTCOMES:
Mouth opening, lateral protrusive movement: will be obtained by a caliper. | Mouth opening, lateral protrusive movement will be measured : 1.day1 before the start of laser therapy, 2.week 1 3. week2 4.week 3 5. week 4 6.one month later 7. 3 months later.
  Mouth opening, lateral protrusive movement: will be obtained by a caliper.

OTHER OUTCOMES:
Clicking: will be obtained by Yes or No. | Clicking will be measured : 1.day1 before the start of laser therapy, 2.week 1 3. week2 4.week 3 5. week 4 6.one month later 7.after 3 months.
  Clicking: will be obtained by Yes or No.
Clicking: will be obtained by Yes or No. | Clicking will be measured : 1.day1 before the start of laser therapy, 2.week 1 3. week2 4.week 3 5. week 4 6.one month later 7. 3 months later.
  Clicking: will be obtained by Yes or No.